CLINICAL TRIAL: NCT04126304
Title: Multi-center Investigation and Study of Mycoplasma Pneumoniae Infection and Macrolide Drug Resistance in Outpatient and In-hospital Pediatric Acute Respiratory Diseases Illness in China
Brief Title: Mycoplasma Infection Rate and Macrolides Resistance in Children With Acute Respiratory Tract Infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Children's Medical Center (Other)
Collaborators: Beijing Children's Hospital (Other); Tianjin Children's Hospital (Other); Xi 'an children's hospital (Unknown); Shenzhen Children's Hospital (Other Government); Third Affiliated Hospital of Zhengzhou University (Other); Shanghai Children's Hospital (Other); Children's Hospital of Chongqing Medical University (Other); Wuhan Children's Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SCMCIRB-K2019060-1
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Respiratory Tract Infections
Keywords: community-acquired pneumonia; common cold; acute bronchitis; Post-infection cough; Mycoplasma infection rate; macrolides resistance
MeSH Terms: conditions — Respiratory Tract Infections; Community-Acquired Pneumonia; Common Cold; Bronchitis | interventions — Azithromycin; Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples Pharyngeal swab Sputum samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Common cold: A cold is a clinical diagnosis.Complaints may include a stuffy nose, sore throat, cough and headache.Objective signs are rare, but may include fever, enlarged anterior cervical lymph nodes, nasal mucosa and oropharyngeal erythema, and nasal mucus.
  Interventions: Drug: Azithromycin; Diagnostic Test: Mycoplasma detection; Other: Data collection
- acute bronchitis: In 2011, the European society of respiratory diseases (ERS) defined acute disease in patients with non-chronic lung disease. Symptoms include cough, with or without expectoration of phlegm, and other symptoms and signs may indicate lower respiratory tract infection and cannot be explained by other diseases (e.g., sinusitis, asthma).The main symptoms of acute bronchitis are cough, may be accompanied by fever, fatigue, asthma and dyspnea.
  Interventions: Drug: Azithromycin; Diagnostic Test: Mycoplasma detection; Other: Data collection
- Post-infection cough: The definition in the 2013 guidelines for diagnosis and treatment of chronic cough in Chinese children: cough refers to a recent history of respiratory tract infection;The cough lasted > for 4 weeks, presenting an irritating dry cough or a little white phlegm.Chest x - ray examination showed no abnormality or only increased lung veins.The pulmonary ventilation function was normal, or presented transient high airway response.Coughs are usually self-limited, and other diagnoses should be considered if the cough is more than 8 weeks old.In addition to other causes of chronic cough.
  Interventions: Drug: Azithromycin; Diagnostic Test: Mycoplasma detection; Other: Data collection
- community-acquired pneumonia: According to the 2019 guidelines for the diagnosis and treatment of community-acquired pneumonia in children, it is defined as infectious pneumonia developed outside the hospital (community), including pneumonia developed after admission due to infection of pathogens with a clear incubation period outside the hospital (community).
  Interventions: Drug: non-macrolides antibiotics; Diagnostic Test: Mycoplasma detection; Other: Data collection

INTERVENTIONS:
Drug: Azithromycin — If the diagnosis is common cold, acute bronchitis or post-infection cough ，treated with non-macrolides when the mycoplasma colloidal gold test is negative, treated with azithromycin when colloidal gold test is positive.
  Groups: Common cold; Post-infection cough; acute bronchitis
Drug: non-macrolides antibiotics — If the diagnosis is community-acquired pneumonia with negative mycoplasma antibody-granule agglutination, non-macrolides are used for treatment
  Groups: community-acquired pneumonia
Diagnostic Test: Mycoplasma detection — 1. common cold, acute bronchitis or post-infection cough :MPlgM colloidal gold detection;Pharyngeal swab MP-RNA PCR, mutated gene detection at 2063 and 2064 site of macrolide-resistant 23S rRNA II region detection
  2. community-acquired pneumonia:mycoplasma antigen antibody particle agglutination detection ;Sputum MP-RNA PCR, mutated gene detection at 2063 and 2064 site of macrolide-resistant 23S rRNA II region detection
Other: Data collection — 1. Common cold:On enrollment, day 3 and day 7, scores were collected based on the Canadian acute respiratory diseases and influenza scale (CARIFS scale), success rate of initial treatment, antimicrobial conversion rate, intravenous rehydration rate, pneumonia conversion rate, re-visit rate, and hospitalization rate.
  2. Acute bronchitis :on enrollment, day 3, and day 7, the Likert 7 subscale was used to score the cough severity questionnaire, collect the success rate of initial treatment, antimicrobial conversion rate, intravenous rehydration rate, pneumonia conversion rate, re-visit rate, and hospitalization rate.
  3. Post-infection cough:on the day after outpatient visit, day 3, day 7, and day 14, the cough severity questionnaire (Likert 7 subscale) was used to score the success rate of initial treatment, antimicrobial conversion rate, intravenous rehydration rate, pneumonia conversion rate, re-visit rate, and hospitalization rate.
  Groups: Common cold; Post-infection cough; acute bronchitis
Other: Data collection — Acquisition of children hospitalized time, heating time, mixed infection, drug (azithromycin, tetracycline, quinolone) dose and use time, pulmonary complication (pleural effusion, atelectasis, necrotizing pneumonia, interstitial pneumonia, occlusive bronchitis, occlusive bronchiolitis, lung, emphysema, lung abscess, bronchiectasis, transparent), pleural puncture/drainage, bronchoscope, oxygen time, into the ICU, mechanical ventilation time, surgery, and deaths and re-visit, hospitalization, surgery and death within 30 days after discharge
  Groups: community-acquired pneumonia

SUMMARY:
In recent years, mycoplasma pneumoniae caused more than 30% of respiratory infections in children in China, among which the detection rate of drug-resistant mycoplasma pneumoniae was higher than 90%. Pediatricians are facing great challenges.

In this study, a total of 2312 clinical cases were expected to be collected, including 1160 cases of outpatient respiratory infection including common cold, acute bronchitis and cough after infection, and 1152 cases of hospitalized community-acquired pneumonia, through uniform enrollment in 11 multi-centers for 1 year. Clinical data and respiratory samples were collected and clinical follow-up was completed.To investigate the infection rate and drug resistance gene of mycoplasma pneumoniae in children's respiratory tract infection.To evaluate the effectiveness of azithromycin in the treatment of mycoplasma pneumoniae respiratory infection.The early prediction model of refractory mycoplasma pneumoniae was established.To explore the clinical value of colloidal gold in early diagnosis of mycoplasma pneumoniae infection

DETAILED DESCRIPTION:
This research center is a cross-sectional investigation and study, 8 centers including Shanghai children's medical center recruit the outpatient respiratory infection cases into the group, 6 centers including Shanghai children's medical recruit children with community-acquired pneumonia in hospital into the group All of the above cases in the group relevant clinical datas are collected, and complete clinical follow-up.Pharyngeal swabs or sputum specimens collected during the study were sent to Shanghai children's medical center for the detection of MP and macrolidene drug resistance genes.

Azithromycin was administered orally or intravenously to outpatients who tested positive for mycoplasma pneumoniae by colloidal gold method.Finally, MP infection rate of children with respiratory diseases including outpatient (common cold, acute bronchitis and cough after infection) and hospitalization (community-acquired pneumonia) was statistically observed.The detection rate of MP macrolides drug resistance gene was isolated from respiratory disease cases.Sensitivity and specificity of MP rapid detection method (antigen and antibody detection rapid colloidal gold method) for diagnosis of MP infection;Effectiveness of azithromycin in treatment of MRMP infection.

ELIGIBILITY:
Inclusion Criteria:

A) age: over 28 days, under 18 years old; B) diagnosis: outpatient diagnosis of common cold, acute bronchitis or post-infection cough and hospitalization cases consistent with community-acquired pneumonia.

C) the guardian of the child (< 8 years old) or the child (≥8 years old) can understand and be willing to participate in this study and sign a written informed consent.

Exclusion Criteria:

A)It is necessary to exclude underlying diseases associated with cardiovascular system, digestive system, nervous system, endocrine system, urinary system, immune system and genetic or chromosomal abnormalities.

B) the children or their families refused to participate in the study.

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The subjects of the study were outpatient patients at 8 centers including Shanghai children's medical center and hospitalized children at 6 centers on Oct. 28, 2019 and Sept. 27, 2020.
Sampling Method: Probability Sample
Enrollment: 2312 (Estimated)
Dates: Start 2019-11-28 (Estimated); Primary Completion 2020-09-27 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
MP infection rates | On enrollment 1 day
  Respiratory illnesses include MP infection rates in children with outpatient (common cold, acute bronchitis, and chronic cough) and hospitalized (community-acquired pneumonia).

SECONDARY OUTCOMES:
MP macrolides drug resistance gene rate | On enrollment 1 day
  The detection rate of MP macrolides drug resistance gene was isolated from respiratory disease cases
Sensitivity and specificity of MP rapid detection method | On enrollment 1 day
  Sensitivity and specificity of MP rapid detection method (antigen and antibody detection rapid colloidal gold method) for diagnosis of MP infection
An early prediction model of refractory MP pneumonia | Community acquired pneumonia 30 days after discharge
  An early prediction model of refractory MP pneumonia caused by MRMP was established
Clinical efficacy of azithromycin | Common cold and acute bronchitis for 7 days ;Post-infection cough for 14 days
  Common cold and acute bronchitis on enrollment, day 3 and day 7;Post-infection cough on the day after outpatient visit, day 3, day 7, and day 14

CONTACTS AND LOCATIONS:
Overall Officials: Yong Yin, master, Principal Investigator — Shanghai Children's Medical Center

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li L, Liao X, Zhao J, Xie YM. [Interpretation of chinese clinical guidelines for acute upper respiratory tract infection in children]. Zhongguo Zhong Yao Za Zhi. 2017 Apr;42(8):1510-1513. doi: 10.19540/j.cnki.cjcmm.2017.0049. Chinese. PMID 29071854
- [Result] Leung DT, Chisti MJ, Pavia AT. Prevention and Control of Childhood Pneumonia and Diarrhea. Pediatr Clin North Am. 2016 Feb;63(1):67-79. doi: 10.1016/j.pcl.2015.08.003. PMID 26613689
- [Result] Nair H, Simoes EA, Rudan I, Gessner BD, Azziz-Baumgartner E, Zhang JSF, Feikin DR, Mackenzie GA, Moiisi JC, Roca A, Baggett HC, Zaman SM, Singleton RJ, Lucero MG, Chandran A, Gentile A, Cohen C, Krishnan A, Bhutta ZA, Arguedas A, Clara AW, Andrade AL, Ope M, Ruvinsky RO, Hortal M, McCracken JP, Madhi SA, Bruce N, Qazi SA, Morris SS, El Arifeen S, Weber MW, Scott JAG, Brooks WA, Breiman RF, Campbell H; Severe Acute Lower Respiratory Infections Working Group. Global and regional burden of hospital admissions for severe acute lower respiratory infections in young children in 2010: a systematic analysis. Lancet. 2013 Apr 20;381(9875):1380-1390. doi: 10.1016/S0140-6736(12)61901-1. Epub 2013 Jan 29. PMID 23369797
- [Result] Basarab M, Macrae MB, Curtis CM. Atypical pneumonia. Curr Opin Pulm Med. 2014 May;20(3):247-51. doi: 10.1097/MCP.0000000000000048. PMID 24626238
- [Result] Blasi F. Atypical pathogens and respiratory tract infections. Eur Respir J. 2004 Jul;24(1):171-81. doi: 10.1183/09031936.04.00135703. PMID 15293621
- [Result] Xu W, Guo L, Dong X, Li X, Zhou P, Ni Q, Zhou X, Wagner AL, Li L. Detection of Viruses and Mycoplasma pneumoniae in Hospitalized Patients with Severe Acute Respiratory Infection in Northern China, 2015-2016. Jpn J Infect Dis. 2018 Mar 22;71(2):134-139. doi: 10.7883/yoken.JJID.2017.412. Epub 2018 Feb 28. PMID 29491245
- [Result] Sondergaard MJ, Friis MB, Hansen DS, Jorgensen IM. Clinical manifestations in infants and children with Mycoplasma pneumoniae infection. PLoS One. 2018 Apr 26;13(4):e0195288. doi: 10.1371/journal.pone.0195288. eCollection 2018. PMID 29698412
- [Result] Wang H, Dai W, Qiu C, Li S, Wang W, Xu J, Li Z, Wang H, Li Y, Yang Z, Feng X, Zhou Q, Han L, Li Y, Zheng Y. Mycoplasma pneumoniae and Streptococcus pneumoniae caused different microbial structure and correlation network in lung microbiota. J Thorac Dis. 2016 Jun;8(6):1316-22. doi: 10.21037/jtd.2016.04.63. PMID 27293852
- [Result] Zhao F, Liu J, Shi W, Huang F, Liu L, Zhao S, Zhang J. Antimicrobial susceptibility and genotyping of Mycoplasma pneumoniae isolates in Beijing, China, from 2014 to 2016. Antimicrob Resist Infect Control. 2019 Jan 24;8:18. doi: 10.1186/s13756-019-0469-7. eCollection 2019. PMID 30697421
- [Result] Yang HJ, Song DJ, Shim JY. Mechanism of resistance acquisition and treatment of macrolide-resistant Mycoplasma pneumoniae pneumonia in children. Korean J Pediatr. 2017 Jun;60(6):167-174. doi: 10.3345/kjp.2017.60.6.167. Epub 2017 Jun 22. PMID 28690643
- [Result] Matsuoka M, Narita M, Okazaki N, Ohya H, Yamazaki T, Ouchi K, Suzuki I, Andoh T, Kenri T, Sasaki Y, Horino A, Shintani M, Arakawa Y, Sasaki T. Characterization and molecular analysis of macrolide-resistant Mycoplasma pneumoniae clinical isolates obtained in Japan. Antimicrob Agents Chemother. 2004 Dec;48(12):4624-30. doi: 10.1128/AAC.48.12.4624-4630.2004. PMID 15561835
- [Result] Bebear C, Pereyre S, Peuchant O. Mycoplasma pneumoniae: susceptibility and resistance to antibiotics. Future Microbiol. 2011 Apr;6(4):423-31. doi: 10.2217/fmb.11.18. PMID 21526943
- [Result] Kawai Y, Miyashita N, Kubo M, Akaike H, Kato A, Nishizawa Y, Saito A, Kondo E, Teranishi H, Wakabayashi T, Ogita S, Tanaka T, Kawasaki K, Nakano T, Terada K, Ouchi K. Nationwide surveillance of macrolide-resistant Mycoplasma pneumoniae infection in pediatric patients. Antimicrob Agents Chemother. 2013 Aug;57(8):4046-9. doi: 10.1128/AAC.00663-13. Epub 2013 May 28. PMID 23716043
- [Result] Yin YD, Wang R, Zhuo C, Wang H, Wang MG, Xie CM, She DY, Yuan X, Wang RT, Cao B, Liu YN. Macrolide-resistant Mycoplasma pneumoniae prevalence and clinical aspects in adult patients with community-acquired pneumonia in China: a prospective multicenter surveillance study. J Thorac Dis. 2017 Oct;9(10):3774-3781. doi: 10.21037/jtd.2017.09.75. PMID 29268385
- [Result] Lee E, Cho HJ, Hong SJ, Lee J, Sung H, Yu J. Prevalence and clinical manifestations of macrolide resistant Mycoplasma pneumoniae pneumonia in Korean children. Korean J Pediatr. 2017 May;60(5):151-157. doi: 10.3345/kjp.2017.60.5.151. Epub 2017 May 31. PMID 28592978
- [Result] Pereyre S, Charron A, Hidalgo-Grass C, Touati A, Moses AE, Nir-Paz R, Bebear C. The spread of Mycoplasma pneumoniae is polyclonal in both an endemic setting in France and in an epidemic setting in Israel. PLoS One. 2012;7(6):e38585. doi: 10.1371/journal.pone.0038585. Epub 2012 Jun 6. PMID 22701675
- [Result] Pereyre S, Touati A, Petitjean-Lecherbonnier J, Charron A, Vabret A, Bebear C. The increased incidence of Mycoplasma pneumoniae in France in 2011 was polyclonal, mainly involving M. pneumoniae type 1 strains. Clin Microbiol Infect. 2013 Apr;19(4):E212-7. doi: 10.1111/1469-0691.12107. Epub 2012 Dec 22. PMID 23279613
- [Result] Yamada M, Buller R, Bledsoe S, Storch GA. Rising rates of macrolide-resistant Mycoplasma pneumoniae in the central United States. Pediatr Infect Dis J. 2012 Apr;31(4):409-0. doi: 10.1097/INF.0b013e318247f3e0. PMID 22209916